CLINICAL TRIAL: NCT02806284
Title: Pneumococci and Hib Vaccination Early and Late After Neurotrauma or Neurosurgery
Brief Title: Pneumococci and Hib Vaccination After Neurotrauma or Neurosurgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPN 00-254
Record Dates: First submitted 2016-05-30; First posted 2016-06-20 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Meningitis
Keywords: vaccination; Streptococcus pneumoniae
MeSH Terms: conditions — Meningitis | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Hiberix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neurotrauma (Active Comparator): Patients with basilar skull fracture with or without known cerebrospinal fluid leakage were enrolled in the neurotrauma (NT) group. All patients were vaccinated with two vaccines at the same time, 0,5 ml PPSV23 and 0,5 ml Act-HIB which is a conjugate vaccine against H. influenzae type b.The vaccines were administered by subcutaneous injections within 10 days from trauma.
  Interventions: Biological: PPSV23, Act-HIB
- Neurosurgery (Active Comparator): Patients scheduled for elective, transsphenoidal pituitary gland surgery were assigned to the neurosurgery (NS) group. All patients were vaccinated with two vaccines at the same time, 0,5 ml PPSV23 and 0,5 ml Act-HIB which is a conjugate vaccine against H. influenzae type b.The vaccines were administered by subcutaneous injections within 10 days from surgery.
  Interventions: Biological: PPSV23, Act-HIB
- Control (Active Comparator): All control patients had undergone neurotrauma with or without basilar skull fracture, or had neurosurgery, at least three weeks earlier. All patients were vaccinated with two vaccines at the same time, 0,5 ml PPSV23 and 0,5 ml Act-HIB which is a conjugate vaccine against H. influenzae type b. They were vaccinated at least three weeks after trauma or surgery. The vaccines were administered by subcutaneous injections.
  Interventions: Biological: PPSV23, Act-HIB

INTERVENTIONS:
Biological: PPSV23, Act-HIB — described in "Arm description"
  Other Names: PPSV23=Pneumovax,

SUMMARY:
The purpose of this study is to determine wether skull trauma or neurosurgery affect the immune response to two vaccine types.

DETAILED DESCRIPTION:
There is a risk of meningitis after neurotrauma and different actions have been taken to reduce this risk. Prophylactic antibiotics are often administered, although at present there is little evidence to support such a regimen. Increasing problems with antibiotic resistance heightens the need for pertinent use of antibiotics.

Even if most of these infections occur early in the course, the risk appears to persist for many years and almost half of the posttraumatic meningitis cases occur after one month. Streptococcus pneumoniae is the most common causative agent and pneumococcal vaccination after neurotrauma is now recommended in several national guidelines. There are, however, no recommendations of when to administer the vaccine. In clinical practice, vaccination is most often performed several weeks after the trauma. Because the risk of meningitis is at the highest shortly after the trauma, vaccination within days would be preferable. Until recently, pneumococcal polysaccharide vaccine (PPSV) was the most common recommendation. During recent years pneumococcal conjugate vaccines (PCV) have been introduced, offering long-term protection and is now recommended in the USA.

Trauma, as well as surgery, activate the innate immune system resulting in, among other things, decreased T-cell function. Patients with injuries of the central nervous system (CNS) may show signs of a specific CNS-injury-induced immune deficiency syndrome (CIDS), which is also characterized by impaired T-cell activity. Accordingly, it can be speculated that ongoing anti-inflammatory response after trauma, here referred to as trauma-induced immune deficiency syndrome (TIDS), and CIDS by impaired T-cell function could negatively affect the response to vaccines, especially to T-cell dependent conjugate vaccines. In the present thesis, focus will be the impact of TIDS and CIDS on the response to T-cell dependent and T-cell independent vaccines.

Methods

Vaccination A conjugate vaccine against Haemophilus influenzae type b (Hib) was chosen as the T-cell-dependent antigen. All patients received a single subcutaneous injection of 0.5 ml Act-HIB® (Sanofi Pasteur MSD, Lyon, France) in the upper right arm. A 0.5 ml dose of this vaccine contains 10 μg of Hib polysaccharide conjugated to 24 micrograms of tetanus protein.

All patients also received, at the same time, a single subcutaneous injection of 0.5 ml Pneumovax® (Sanofi Pasteur MSD AB, Lyon, France) (PPSV23) containing 25 μg of purified capsular polysaccharide from each of the 23 serotypes (1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F and 33F) in the upper left arm.

Patients in the NT and NS groups were vaccinated within 10 days after trauma or surgery. Control patients were vaccinated, according to the local routine for pneumococcal vaccination, at least three weeks after trauma or surgery.

Adverse reactions to the vaccine were recorded in the case report form.

Sera collection and analysis Pre-vaccination sera were collected just before vaccination and post-vaccination sera were obtained three and six weeks after vaccination. Samples were stored at -70oC pending analysis. The laboratory was blinded with respect to group assignment of the patients.

IgG antibody concentrations to Hib polysaccharide were determined by enzyme immunoassay which is an established and accredited methodology.

An anti-Hib polysaccharide antibody concentration of 0.15 -1.0 μg/ml has been associated with long-term protection against invasive Hib infection after vaccination of children with Hib polysaccharide vaccine. Based on previous experience in children, a post-vaccination concentration of 10 μg/ml, 10 times the upper supposed protective concentration, was chosen as the target level for a good response to the vaccination in this study.

Serotype-specific anti-polysaccharide binding IgG antibody levels to serotypes 4, 6B, 9V, 14, 18C, 19F and 23F were determined by enzyme immunoassay which is an established and accredited methodology.

A serotype-specific IgG >0.35 μg/ml has been defined as the correlate of protection for invasive disease in infant recipients of (PCV). The true correlate of protection for adults after vaccination with PPSV23 is not known. The value of 1.0 μg/ml was chosen as the target level for a good response to the vaccination in this study.

ELIGIBILITY:
Inclusion Criteria:

* Basilar skull fracture or transsphenoidal pituitary gland surgery
* Own or presumed consent (by next of kin of unconscious)

Exclusion criteria

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2001-01; Primary Completion 2008-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of IgG anti-Hib (ug/ml) | baseline and 3 weeks
Change from baseline of IgG anti-Hib (ug/ml) | baseline and 6 weeks
Change from baseline of specific IgG against pneumococcal serotypes 4, 6B, 9V, 14, 18C, 19F and 23F (ug/ml) | baseline and 3 weeks
Change from baseline of specific IgG against pneumococcal serotypes 4, 6B, 9V, 14, 18C, 19F and 23F (ug/ml) | baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sjölin, Professor, Principal Investigator — Uppsala University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hedberg AL, Pauksens K, Enblad P, Soderberg J, Johansson B, Kayhty H, Sjolin J. Pneumococcal polysaccharide vaccination administered early after neurotrauma or neurosurgery. Vaccine. 2017 Feb 7;35(6):909-915. doi: 10.1016/j.vaccine.2016.12.065. Epub 2017 Jan 6. PMID 28069358